CLINICAL TRIAL: NCT00531466
Title: AV650-014: A Four Week, Prospective, Randomized, Double Blind, Placebo-Controlled Trial to Assess Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of AV650 in Patients With Spasticity Due to Spinal Cord Injury
Brief Title: Safety and Preliminary Effectiveness of AV650 in Patients With Spasticity Due to Spinal Cord Injury
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Avigen (Industry)
Responsible Party: Robert Elfont, MD, Avigen, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AV650-014
Record Dates: First submitted 2007-09-14; First posted 2007-09-18 (Estimated); Last update posted 2008-11-04 (Estimated); Status verified 2008-11

CONDITIONS: Muscle Spasticity
Keywords: Spinal cord injury
MeSH Terms: conditions — Muscle Spasticity; Spinal Cord Injuries | interventions — Tolperisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: tolperisone HCl (AV650)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tolperisone HCl (AV650) — One tablet orally three times a day for 28 days
  Arms: 1
Drug: Placebo — One tablet orally three times a day for 28 days
  Arms: 2

SUMMARY:
A drug called AV650 (tolperisone HCl) will be given to patients who have spasticity following a spinal cord injury. This study has three purposes:

1. To determine whether AV650 is safe for patients with spinal cord injury;
2. To assess what the body does with AV650 once it is ingested; and,
3. To gather some early evidence as to whether AV650 is effective in treating spasticity in patients with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who provide written informed consent.
* Male or female subjects aged 18 to 70 years.
* In the judgment of the Principal Investigator, able to comply with protocol requirements.
* Subjects willing and able to withdraw from other anti-spasmodic/muscle relaxant drugs for at least two weeks before randomization (including but not limited to baclofen, benzodiazepines, clonazepam, clonidine, dantrolene, diazepam, gabapentin, and tizanidine).
* Neurological level between C-4 and T-12 spinal cord levels.
* SCI duration of 6 or more months.
* Muscle tone sufficient to score at least two (2) on the Ashworth Scale for at least one of the following lower muscle groups: ankle plantar flexors (gastrocnemius), knee extensors (quadriceps), knee flexors (hamstrings) and/or hip adductors (adductors) and seven (7) for the most spastic limb.
* ASIA Impairment Scale Exam score of B, C or D.
* Female subjects of childbearing potential must be either surgically sterile or using an effective method of contraception.
* Female subjects of childbearing potential must have a negative urine pregnancy test at baseline (Study Day 0).

Exclusion Criteria:

* Subjects with a known hypersensitivity to lidocaine or non-steroidal analgesics.
* Subjects with clinically significant cardiovascular, pulmonary, endocrine, hepatic, renal, neurological, metabolic, or psychiatric disease.
* Any recent history of mental illness, drug addiction, recreational drug use, or alcoholism and/or any similar condition that the investigator feels should prohibit study participation.
* Any significant illness during the four weeks preceding Study Day 1.
* History of cancer or inflammatory arthritis of large joints.
* History of gastric or duodenal ulcer.
* Concurrent symptomatic urinary tract infections with fever.
* Severe physical injury, direct impact trauma, or neurological trauma within the last 6 months not including Spinal Cord Injury.
* ASIA Impairment Scale score of A or E.
* Uncontrolled hypertension or hypotension.
* Percussive tenderness of vertebral body or spinous process.
* Subjects with corrective surgery to or contracture of the measurable hip, knee, or ankle joints.
* Subjects known to be Hepatitis B or HIV positive.
* Female subjects who are pregnant or nursing.
* Subjects who have received an investigational drug within 30 days before Screening visit.
* Subjects with any documented episodes of seizures.
* Subjects requiring use of clinically relevant 2C19 or 2D6 inhibitors, or concomitant use of lidocaine.
* Use of rescue medication(s) within 48 hours of baseline procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To assess the safety, tolerability and PK profile of AV650 in subjects with spasticity due to spinal cord injury. | 1 month

SECONDARY OUTCOMES:
To determine preliminary efficacy in subjects with spasticity due to SCI | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ralph J Marino, MD, Principal Investigator — Thomas Jefferson University
Locations (10):
- United States (9):
  - Southern California Clinical Research, Inc., Pasadena, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Shepherd Center, Inc., Atlanta, Georgia
  - Internal Center for Spinal Cord Injury Kennedy Kreiger Institute, Baltimore, Maryland
  - Kernan Orthopaedics & Rehab. Hospital, Baltimore, Maryland
  - Kessler Institute for Rehab., West Orange, New Jersey
  - Carolinas Rehabilitation, Charlotte, North Carolina
  - Jefferson Medical College of Thomas Jefferson University, Philadelphia, Pennsylvania
  - Hunter Holmes McGuire Veterans Affairs Medical Center, Richmond, Virginia
- Rehabilitation Hospital Health Sciences Centre, Winnipeg, Quebec, Canada